CLINICAL TRIAL: NCT06545786
Title: Intraoperative Diagnosis of Neurocognitive Complications Via Electroencephalographic (IDEA Network)
Brief Title: Intraoperative Diagnosis of Neurocognitive Complications Via Electroencephalographic Analysis
Status: Recruiting | Type: Observational
Sponsor: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, PhD, Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Other Study IDs: IDEA Network
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Surgery; Postoperative Delirium; Anesthesia; Silent Stroke; Emergence Delirium
Keywords: Non-cardiac surgery; Anesthesia; Postoperative Delirium; Silent Stroke; Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-cardiac surgery: Patients scheduled for non-cardiac surgery of intermediate to high risk
  Interventions: Device: Intraoperative electroencephalography

INTERVENTIONS:
Device: Intraoperative electroencephalography — EEG recording will be performed using the standard 16-electrode configuration according to the international "10-20" system. During the recording, electrode impedances will be maintained at a level not exceeding 5 kilo-ohms.

SUMMARY:
Postoperative neurocognitive disorders (PND) are serious and common complications after surgery, especially in elderly patients. These disorders can affect cognitive functions for years, deteriorating quality of life and increasing hospital stays and medical costs. Diagnosing PND is challenging due to their varied manifestations, such as memory and attention problems, and the lack of standardized criteria and biomarkers.

One well-studied form of PND is postoperative delirium (POD). According to the ICD-10, POD is an organic cerebral syndrome characterized by disturbances in consciousness, attention, perception, and other cognitive functions. Researchers suggest that POD development involves a combination of predisposing and precipitating factors.

Electroencephalography (EEG) has been used in anesthesiology to assess anesthesia depth and intraoperative awareness. Modern EEG analysis methods, like spectral analysis, offer new ways to evaluate patients' neurophysiological states. Studies show that EEG monitoring can predict complications such as intraoperative stroke and delirium, particularly in cardiothoracic and neurosurgical operations.

The relationship between EEG patterns and POD is not well understood. Specific EEG patterns may indicate the risk of POD, aiding in the identification of risk factors and prevention methods. This could help anesthesiologists and surgeons optimize their approaches, reducing the risk of cognitive complications.

DETAILED DESCRIPTION:
Postoperative Neurocognitive Disorders (PND) are one of the most serious and common complications following surgery, especially in elderly patients. Postoperative neurocognitive disorders can impact cognitive functions for a prolonged period post-surgery, sometimes lasting several years. This not only deteriorates the quality of life but also increases hospitalization time and medical costs.

The difficulty in diagnosing postoperative neurocognitive disorders is that postoperative neurocognitive disorders can manifest in various forms, including memory, attention, and executive function problems. The lack of standardized diagnostic criteria and clear biomarkers complicates early identification and prognosis of postoperative neurocognitive disorders.

One of the most studied forms of postoperative neurocognitive disorders is postoperative delirium (POD). Currently, the concept of postoperative delirium development suggests a combination of predisposing and precipitating factors. Furthermore, according to the ICD-10, postoperative delirium is defined as an etiologically nonspecific organic cerebral syndrome characterized by disturbances in consciousness, attention, perception, thinking, memory, psychomotor behavior, emotions, and the sleep-wake cycle. The indication of an organic nature of the lesion prompts researchers to explore the possibility of diagnosing brain dysfunctions clinically manifesting as postoperative delirium.

Electroencephalography (EEG) has long been used in anesthesiology to assess the depth of anesthesia and the risk of awareness during surgery. With the use of modern analysis algorithms, such as spectral analysis and synchronization between different brain regions, electroencephalography opens new horizons for assessing the patient's neurophysiological state. Currently, the use of electroencephalography for monitoring cerebral perfusion and oxygenation is being studied, which is especially critical during cardiothoracic and neurosurgical operations. One study showed that a new interhemispheric similarity index in electroencephalography could serve as an indicator of the risk of complications such as intraoperative stroke and delirium after cardiac surgery. These data demonstrate the possibility of using electroencephalography monitoring as a tool for predicting adverse neurocognitive outcomes.

The relationship between electroencephalography and postoperative delirium has not been sufficiently studied. The hypothesis is that specific electroencephalography patterns may serve as indicators of the organic substrate development of postoperative delirium, which may lead to the study of risk factors and methods of their prevention. This, in turn, will allow anesthesiologists and surgeons to optimize approaches to anesthesia and surgical intervention, minimizing the risk of negative cognitive consequences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled non-cardiac surgery of intermediate or high risk
* General anesthesia using inhalational anesthetics
* Informed consent from the patient to participate in the study

Exclusion Criteria:

* Preoperative MMSE score less than 20 points
* History of any mental illness
* Use of psychotropic drugs within 1 month prior to inclusion in the study
* Presence of neuromuscular diseases
* Neurosurgical procedures
* Inability to undergo preoperative testing for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for non-cardiac surgery of intermediate to high risk
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of mean intraoperative alpha rhythm power for the development of postoperative delirium | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
Prognostic value of mean intraoperative alpha rhythm power for the development of early postoperative neurocognitive disorders | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
Prognostic value of mean intraoperative alpha rhythm power for the development of intraoperative silent brain infarction | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.

SECONDARY OUTCOMES:
Prognostic value of maximum intraoperative alpha rhythm power for the development of postoperative delirium | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
Prognostic value of maximum intraoperative alpha rhythm power for the development of early postoperative neurocognitive disorders | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
Prognostic value of maximum intraoperative alpha rhythm power for the development of silent brain infarction | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
The prognostic capability of the "burst suppression" pattern for predicting the development of silent brain infarction | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
The prognostic capability of the "burst suppression" pattern for predicting the development of postoperative delirium. | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
The prognostic capability of the "burst suppression" pattern for predicting the development of early postoperative neurocognitive disorders. | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
The prognostic value of early postoperative neurocognitive disorders for predicting the development of postoperative delirium. | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
The prognostic value of postoperative delirium for predicting the development of silent brain infarction | Through study completion, an average of 3 year
  The prognostic value assessment is performed using the area under the ROC curve (AUROC). The value ranges from 0.5 to 1.0. The closer the AUROC value is to one, the higher the prognostic capability of the electroencephalography.
28-days mortality | 28 days
  Number of deaths in period of 28 days after enrollment
1-year mortality | 1 year
  Number of deaths in period of 1 year after enrollment

OTHER OUTCOMES:
Serum level of S100 beta protein | within 1 hour before surgery, 1 hour after surgery
Serum level of Interleukin-6 | within 1 hour before surgery, 1 hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, PhD, Principal Investigator — Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Locations (1):
- City clinical hospital named after SS Yudin, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No